CLINICAL TRIAL: NCT00941772
Title: Confirmation of Nasogastric Tube Placement Via Ultrasonography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oklahoma State University Center for Health Sciences (Other)
Responsible Party: Bryan Menges D.O., OklahomaSU
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2008017
Record Dates: First submitted 2009-07-06; First posted 2009-07-20 (Estimated); Last update posted 2010-12-02 (Estimated); Status verified 2010-12

CONDITIONS: Nasogastric Tube Intubation
Keywords: Nasogastric tube verification with ultrasonography; ultrasonography
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Ultrasonography — Verify nasogastric tube placement with ultrasonography and compare its accuracy with plain radiography

SUMMARY:
The purpose of the study is to determine if ultrasonography is an adequate means for confirmation of nasogastric tube placement and that ultrasonography is more time efficient than radiography confirming nasogastric tube placement.

DETAILED DESCRIPTION:
Our current nasogastric tube placement protocol requires confirmation of nasogastric tube placement with plain radiography. Obtaining a plane radiograph in the emergency department can be time consuming and exposes the patient to radiation. Ultrasound is readily available to our physicians and does not expose patients to radiation.

Confirmation of nasogastric tube placement by ultrasonography may provide a faster means of confirmation and expose patients to less radiation.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female Patients 18 years of age or older.
* Patients in the emergency department at Oklahoma State University Medical Center that require NG intubation with radiography confirmation.

Exclusion Criteria:

* Patients under the age of 18 years of age.
* Patients that are prisoners of the State or Government.
* Patient is pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-02 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Ultrasonography is as accurate as plain radiograph in confirming nasogastric tube placement | one year

CONTACTS AND LOCATIONS:
Overall Officials: Bryan J Menges, D.O., Principal Investigator — Oklahoma State University of Health Sciences
Locations (1):
- Oklahoma State University Medical Center, Tulsa, Oklahoma, United States